CLINICAL TRIAL: NCT03327922
Title: Interrupted Subdermal Suture Spacing During Linear Wound Closures and the Effect on Wound Cosmesis: a Randomized Evaluator Blinded Split Wound Comparative Effectiveness Trial
Brief Title: Interrupted Subdermal Suture Spacing During Linear Wound Closures and the Effect on Wound Cosmesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 1115591
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Interrupted Subdermal Suture
Keywords: Subdermal; Suture; Wound Closure; Wound Cosmesis

STUDY DESIGN:
Intervention Model Description: At the follow-up visit, two blinded observers will record their scores independently using the physician observer scar assessment score instrument (POSAS).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Vicryl absorbable suture placed 2 cm apart (Experimental): Wound closed with sutures spaced 2 centimeters apart will be treated in a simple, interrupted subdermal suture pattern
  Interventions: Device: Vicryl absorbable suture
- Vicryl absorbable suture placed 1 cm apart (Experimental): Wound closed with sutures spaced 1 centimeter apart will be treated in a simple, interrupted subdermal suture pattern
  Interventions: Device: Vicryl absorbable suture

INTERVENTIONS:
Device: Vicryl absorbable suture — Vicryl absorbable suture is a synthetic sterile surgical suture made up of a copolymer

SUMMARY:
This study aims to investigate whether the spacing of the interrupted deep (subdermal) sutures affects surgical wound cosmesis on the trunk and extremities. In other words, the investigator would like to determine which of the following yields a more cosmetically appealing scar: many closely approximated subdermal sutures or fewer, more widely spaced subdermal sutures. The investigator wishes to compare the effects of one versus two centimeter spacing between sutures.

DETAILED DESCRIPTION:
Sutures are the standard of care in repairing cutaneous wounds. The majority of surgical reconstructions following a Mohs micrographic surgery and standard surgical excisions require two layers of sutures: a deep layer and a top layer. The deep layer dissolves naturally whereas the top layer must be removed.

This study aims to investigate whether the spacing of the interrupted deep (subdermal) sutures affects surgical wound cosmesis on the trunk and extremities. In other words, the investigator would like to determine which of the following yields a more cosmetically appealing scar: many closely approximated subdermal sutures or fewer, more widely spaced subdermal sutures. The investigator wishes to compare the effects of one versus two centimeter spacing between sutures. It is possible that fewer, more widely spaced sutures may leave more open space in the wound, leaving more tension to pull on those few sutures, possibly encouraging the wound to dehisce and make it harder to approximate the wound edges yielding a less cosmetically appealing scar compared to placing many closely approximated sutures which would decrease the tension and likely better approximate the wound edges yielding a more cosmetically appealing scar. On the other hand, we may find that suture spacing has no effect on wound cosmesis and that placing fewer, more widely spaced sutures is much more time efficient. The investigator may also find that the effect of suture spacing on wound cosmesis is dependent on wound tension. For example, perhaps the suture pacing would have no effect on the cosmesis of a wound under no tension, however, for a wound under high tension, it is possible that many closely approximated sutures would yield better cosmetic results for the reasons listed above.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the trunk and extremities with predicted primary closure
* Willing to return for follow up visit.

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 4 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Scar Assessment | 3 months following procedure
  The primary endpoint will be the score of two blinded reviewers using the patient observer scar assessment score.

SECONDARY OUTCOMES:
Width of Scar | 3 months following procedure
  A secondary endpoint will include the width of the scar 1 cm from midline on each side
Erythema | 3 months following procedure
  If one half of the scar has more associated erythema, this will be noted

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eshagh K, Sklar LR, Pourang A, Armstrong AW, Dhaliwal H, Eisen DB. Interrupted subcuticular suture spacing during linear wound closures and the effect on wound cosmesis: a randomized evaluator-blinded split-wound comparative effectiveness trial. Br J Dermatol. 2022 Sep;187(3):318-323. doi: 10.1111/bjd.21625. Epub 2022 Jun 13. PMID 35474448